CLINICAL TRIAL: NCT05100316
Title: A Screening Protocol to Support Preliminary Eligibility for Clinical Trials Evaluating Safety and Efficacy of Adoptive Cell Therapies in Participants With Solid Tumors and Hematologic Malignancies
Brief Title: Screening Protocol for Preliminary Eligibility Determination for Adoptive Cell Therapy Trials
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial terminated due to feasibility reasons
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 213033
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-05

CONDITIONS: Neoplasms
Keywords: Adoptive T-cell therapy; Hematologic Malignancy; Human leukocyte antigen; Screening study; Solid Tumors; T-cell receptors
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with solid tumors and hematological malignancies (Other): Participants with solid tumors and hematological malignancies will be included. No study treatment will be administered in this study.
  Interventions: Other: Screening Platform

INTERVENTIONS:
Other: Screening Platform — Eligible participants who qualify as per this screening protocol may be referred to evaluate adoptive cell therapy in participants with various malignancies, on a separate treatment trial. No study treatment will be administered in this screening study.

SUMMARY:
This screening study is intended to determine preliminary eligibility of participants who may be potential candidates for GlaxoSmithKline's Adoptive T-cell therapy studies by screening for appropriate biomarkers. No treatment intervention will occur as part of this screening study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of locally advanced high-risk eligible tumor types .
* Participant must be greater than or equal to (>=)18 years of age (or >=10 years of age with synovial sarcoma or myxoid/round cell liposarcoma [MRCLS])
* Participants with life expectancy of greater than 6 months
* Performance status: Eastern Cooperative Oncology Group 0-1.

Exclusion Criteria:

* Any prior treatment with oncology cell and/or gene therapy (unless agreed in advance with Sponsor)
* Prior malignancy not in complete remission.
* Clinically significant systemic illness
* Serious active infections or significant cardiac, pulmonary, hepatic or other organ dysfunction,
* Prior or active demyelinating disease
* Previous New-York Esophageal Antigen-1 (NY-ESO-1)-specific T cells, NY-ESO-1 vaccine, or NY-ESO-1 targeting antibody.
* Previous allogeneic hematopoietic stem cell transplant within the last 5 years or solid organ transplant.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Waterloo, Iowa
  - GSK Investigational Site, Springfield, Missouri

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This screening study was intended to determine potential eligibility of participants for GlaxoSmithKline's Adoptive T-cell therapy studies by screening for appropriate biomarkers. The study was terminated early due to feasibility reasons.
Pre-assignment Details: A total of 16 participants were enrolled in the study and provided blood sample for biomarker assessment.
Groups:
- Participants With Non-small Cell Lung Cancer (NSCLC): Participants with NSCLC were screened for appropriate biomarkers for an intended adoptive cell therapy on a separate treatment trial. No study treatment was administered in this study.
Period: Overall Study
Arm/Group | Participants With Non-small Cell Lung Cancer (NSCLC)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Non-small Cell Lung Cancer (NSCLC)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.8 (7.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN - JAPANESE HERITAGE | 1
  BLACK OR AFRICAN AMERICAN | 2
  WHITE-WHITE/CAUCASIAN/EUROPEAN HERITAGE | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Human Leukocyte Antigen (HLA) A Genotypes Status
Description: Blood samples were collected for HLA compatibility testing. Number of participants with eligible human leukocyte antigen (HLA) A genotypes status are presented. Data has been reported for following categories: One HLA Allele Positive, Two HLA Allele Positive, Negative and Ambiguous.
Time Frame: Up to 2 weeks
Population: Enrolled population included all participants who provided sample for biomarker assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Non-small Cell Lung Cancer (NSCLC)
Number analyzed (Participants) | 16
Participants
  One HLA Allele Positive | 9
  Two HLA Allele Positive | 1
  Negative | 6
  Ambiguous | 0

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to 2 weeks
Description: Enrolled population was used to assess all-cause mortality, non-SAEs and SAEs which included all participants who provided sample for biomarker assessment.
Arm/Group | Participants With Non-small Cell Lung Cancer (NSCLC)
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT05100316/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT05100316/SAP_001.pdf